CLINICAL TRIAL: NCT05727618
Title: The Effect of Pituitrin on Postoperative Outcomes in Patients With Pulmonary Hypertension Undergoing Cardiac Surgery: a Randomized Controlled Study
Brief Title: The Effect of Pituitrin on the Patients With Pulmonary Hypertension Undergoing Cardiac Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical research protocol failed to obtain approval from the Institutional Review Board (IRB).
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Meng Lv, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LM-KLC-2022
Record Dates: First submitted 2023-01-16; First posted 2023-02-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery; Hypertension, Pulmonary
Keywords: cardiac surgery; Hypertension, Pulmonary; Pituitary Hormones, Posterior; Extracorporeal Circulation
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Pituitary Hormones, Posterior; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pituitrin group (Experimental): The specification of posterior pituitary injection is 1ml/6U, diluted with normal saline to 0.5u/ml, and injected by intravenous pump at the rate of 0.04u/ (kg · h).
  Interventions: Drug: Pituitrin
- normal saline group (Placebo Comparator): Intravenous infusion of normal saline at the same dose and speed
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Pituitrin — The specification of posterior pituitary injection is 1ml/6U, diluted with normal saline to 0.5u/ml, and injected by intravenous pump at the rate of 0.04u/ (kg · h).
  Arms: pituitrin group
Drug: normal saline — Intravenous infusion of normal saline at the same dose and speed
  Arms: normal saline group

SUMMARY:
This study is a parallel group, single blind, randomized controlled trial. Patients with pulmonary hypertension who met the inclusion criteria and planned to undergo elective cardiac surgery under cardiopulmonary bypass from July 1, 2022 to December 1, 2024 in the Department of cardiac surgery of the First Affiliated Hospital of Shandong First Medical University were selected. After removing the aortic blocking forceps, the experimental group immediately injected the test drug (pituitrin 0.04u/ (kg · h)) intravenously, The control group was immediately injected with the corresponding dose of normal saline by intravenous pump. The main outcome was the composite endpoint of all-cause mortality 30 days after operation or common complications after cardiac surgery (stroke, requiring mechanical ventilation for more than 48 hours, deep sternal wound infection, cardiac reoperation, extracorporeal membrane oxygenation, atrial fibrillation or acute renal injury).

DETAILED DESCRIPTION:
Cardiac surgery is the most important treatment for serious coronary heart disease, valvular heart disease, congenital heart disease and other heart diseases. Its postoperative mortality and serious complications have also been widely concerned, especially in patients with pulmonary hypertension. The persistent pulmonary hypertension and systemic vascular paralysis during the perioperative period are the main causes of early postoperative death and serious complications such as organ failure.Catecholamine vasoactive drugs commonly used in cardiac surgery may aggravate the condition of pulmonary hypertension, while the use of drugs to reduce pulmonary hypertension, such as nitric oxide, prostaglandins and phosphodiesterase inhibitors, may worsen the state of systemic vascular paralysis.

Vasopressin and oxytocin are two effective components in pituitrin, and vasopressin is the main component that exerts strong vasoconstrictive effect.Vasopressin binds to receptors distributed in vascular smooth muscle, pituitary and kidney, and exerts its effects by regulating adenosine triphosphate sensitive K+ channel function, nitric oxide production and enhancing vascular response to catecholamine.In addition, oxytocin can also bind to the receptors distributed in the heart and vascular endothelium, and play a role by releasing atrial natriuretic peptide and nitric oxide.Therefore, pituitrin can not only constrict systemic circulation vessels and increase systemic circulation pressure, reduce pulmonary artery pressure and pulmonary vascular resistance, but also protect the heart and kidney.

Therefore, this study intends to explore whether pituitrin has an impact on the prognosis of patients with pulmonary hypertension after cardiac surgery, so as to provide reference for its clinical application.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years and ≤80 years;
* scheduled for elective cardiopulmonary bypass heart surgery (adult congenital heart disease surgery, coronary artery bypass grafting, valve replacement, valvuloplasty, heart transplantation and aortic surgery);
* Patients who had pulmonary hypertension (Mean pulmonary artery pressure at rest ≥ 25mmhg or pulmonary artery systolic pressure (PASP) ≥ 40mmhg as shown by echocardiography);
* sign informed consent.

Exclusion Criteria:

* use pituitrin or vasopressin before operation;
* Patients who had acute coronary syndrome;
* preoperative use of left ventricular assist devices other than intra aortic balloon - pump (IABP);
* Patients who had liver, thyroid and adrenal diseases, severe lung diseases, diabetes;
* Patients who had preoperative renal insufficiency (The increase of serum creatinine (SCR) within 48 h ≥ 0.3mg/dl (or ≥ 26.5 μ mol/L)； Or it is known or speculated that the increase of SCR in the past 7 days is more than 1.5 times of the basic value; Or 0.5ml/kg urine volume per hour for 6H);
* Patients who had severe carotid artery stenosis, preoperative stroke, mental disorder and other difficult to communicate and cooperate;
* Patients who had peripheral vascular disease, allergy to vasopressin or pituitrin, severe hyponatremia (na+ < 130 mmol/l), acute mesenteric ischemia, pregnancy, malignant tumors, required ECMO and underwent emergency surgery or reoperation;
* Patients who had participated in other clinical studies in recent 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
a composite endpoint of mortality or severe postoperative complications | Within 30 days after cardiac surgery
  severe complications after cardiac surgery, including stroke, requirement of mechanical ventilation for longer than 48h, deep sternal wound infection, reoperation, or acute renal failure

SECONDARY OUTCOMES:
incidence of postoperative infection | Within 30 days after cardiac surgery
  The patient appears infection after surgery.
septic shock | Within 30 days after cardiac surgery
  Septic shock was defined as the septic syndrome with shock caused by microorganisms and their toxins.
duration of mechanical ventilation | Time from the beginning of mechanical ventilation to the end of mechanical ventilation up to 30 days after cardiac surgery.
  Total duration of mechanical ventilation during or after surgery.
postoperative pulmonary complications | Within 30 days after cardiac surgery
  This is a composite endpoint indicator, includs atelectasis, pleural effusion, diaphragmatic dysfunction, prolonged mechanical ventilation, pneumonia, pneumothorax, acute respiratory distress syndrome, etc.The occurrence of any of the above pulmonary complications is considered as a positive outcome.
time to achieve hemodynamic stability | Within 30 days after cardiac surgery
  From hemodynamic change to hemodynamic stability.
use of dobutamine or other vasoactive drugs | Within 30 days after cardiac surgery
  The patients use dobutamine or other vasoactive drugs.
incidence of digital ischemia | Within 30 days after cardiac surgery
  Digital ischemia is a symptom caused by insufficient blood supply to the fingers.
acute mesenteric ischemia | Within 30 days after cardiac surgery
  Acute mesenteric ischemia includes arterial and venous thrombosis, thrombosis, and vasoconstriction secondary to low blood flow. Arterial lesions mainly included superior mesenteric artery embolism, superior mesenteric artery thrombosis and non occlusive mesenteric ischemia. The main venous lesions were mesenteric venous thrombosis.
gastrointestinal complications | Within 30 days after cardiac surgery
  Including dyspepsia, abdominal distension, constipation, postoperative stress ulcer, gastrointestinal bleeding, etc.
incidence of acute myocardial infarction | Within 30 days after cardiac surgery
  Acute myocardial infarction is myocardial necrosis caused by acute and persistent ischemia and hypoxia of coronary artery.
new onset tachyarrhythmia | Within 30 days after cardiac surgery
  Tachyarrhythmia includes premature beat, tachycardia, atrial fibrillation and ventricular fibrillation, etc.
water poisoning | Within 30 days after cardiac surgery
  Water poisoning refers to that when the total amount of water ingested by the body greatly exceeds the amount of water discharged, so that water is retained in the body, resulting in the decrease of plasma osmotic pressure and the increase of circulating blood volume.
vasodilative shock | Within 30 days after cardiac surgery
  Vasodilative shock is caused by vasodilation, increased vascular bed volume and relatively insufficient intravascular blood volume, including septic shock, anaphylactic shock and neurogenic shock.
incidence of pulmonary embolism | Within 30 days after cardiac surgery
  Pulmonary embolismwas defined as clinical pathophysiological syndrome of pulmonary circulatory dysfunction caused by pulmonary artery and its branches blocked by various emboli falling off of systemic circulation.
low cardiac output syndrome | Within 30 days after cardiac surgery
  Low cardiac output syndrome refers to the complex pathophysiological changes of insufficient perfusion of multiple organs and tissue hypoxia due to the decrease of cardiac output.
acute respiratory distress syndrome | Within 30 days after cardiac surgery
  Acute respiratory distress syndrome (ARDS) is a clinical syndrome characterized by refractory hypoxemia, which is caused by intrapulmonary and / or extrapulmonary causes.
delirium | Within 30 days after cardiac surgery
  Delirium refers to a group of syndromes, also known as acute brain syndrome. It is manifested as consciousness disorder, disorganized behavior, no purpose and unable to concentrate.
need for renal replacement therapy (RRT) | Within 30 days after cardiac surgery
  Replacement therapy usually includes hemodialysis, peritoneal dialysis and kidney transplantation.
need for hemodialysis | Within 30 days after cardiac surgery
  Hemodialysis (hd) is one of the renal replacement therapies for patients with acute and chronic renal failure.
incidence of readmission to ICU | Within 30 days after cardiac surgery
  The patients re-enters ICU.
length of ICU stay | Within 30 days after cardiac surgery
  From the day of surgery to the time the patient leaves the ICU.
length of stay | Within 30 days after cardiac surgery
  From the day of surgery to the time the patient leaves the hospital.
levels of serum antidiuretic hormone in patients | at entering the operating room(T1), 4 hour(T2), 12 hour(T3) and 24 hour(T4) postoperatively
  T1-T4 were defined as entering the operating room, 4, 12 and 24 hour postoperatively, respectively.
levels of copeptin in patients | at entering the operating room(T1), 4 hour(T2), 12 hour(T3) and 24 hour(T4) postoperatively
  T1-T4 were defined as entering the operating room, 4, 12 and 24 hour postoperatively, respectively.
secondary endotracheal intubation | Within 30 days after cardiac surgery
  Secondary endotracheal intubation refers to the second endotracheal intubation after the patient's postoperative endotracheal intubation is removed.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Li, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University; Meng Lv, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No